CLINICAL TRIAL: NCT04118244
Title: Development of a Functional Test to Assess Fluid Status During Lung Protective Ventilation Strategies in the Operating Room.
Brief Title: A Functional Test to Assess Fluid Status During Lung Protective Ventilation Strategies
Status: Completed | Type: Observational
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jun joohyun, Assistant Professor, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: 2019-07-004-002
Record Dates: First submitted 2019-10-02; First posted 2019-10-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Patients Receiving Protective Lung Ventilation; Patients in Grey Zone (3 < Pulse Pressure Variation (PPV) < 17

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: lung recruitment maneuver — The ventilator was switched to pressure control ventilation, inspiratory time was increased to 50%, the peak inspiratory pressure gradient (above PEEP) was set at 15cm H2O, and PEEP was progressively increased to obtain a stepwise increase of peak inspiratory to 20, 25, and 30 cm H2O every three breaths. The final recruiting pressure of 30 cm H2O was applied for six breaths.

SUMMARY:
Dynamic preload indices, such as pulse pressure variation (PPV) and stroke volume variation (SVV) are generally accepted as accurate indicator of fluid responsiveness in mechanically ventilated patients. Because SVV and PPV are generated by the pressure transmitted from the airways to the pleural and pericardial spaces, their reliability is limited in patients receiving low tidal volume (VT) ventilation and in those with a driving pressure lower than 20 cm H2O.

Lung-protective ventilation using low VT with positive end expiratory pressure (PEEP) has recently been demonstrated to significantly improve postoperative outcome, and its application is gradually increasing in surgical patients. However, protective ventilation alters the predictability of dynamic preload indices and thus limits their use in the operating theatre.

Lung recruitment maneuvers (LRMs), used to reopen collapsed lung, and PEEP have been proposed as the key components of lung-protective ventilation strategy. LRM increases intrathoracic pressure, which in turn causes a transient decrease in stroke volume (SV) and arterial pressure; this may depend on preload status. Interestingly, recent study reported that the augmented PPV during LRM using vital capacity maneuver (VCM, continuous positive airway pressure of 30 cm H2O for 10 s) could predict preload responsiveness under open chest condition.

Investigators hypothesized that the augmented PPV and SVV by a stepwise LRM with incremental PEEP could represent a functional test to suggest preload responsiveness and, therefore, predict fluid responsiveness. The aims of the current study were (1) to assess the ability of augmented PPV and SVV during stepwise LRM-induced to predict fluid responsiveness in mechanically ventilated patients in the operating room, (2) to assess the ability of stepwise LRM-induced decrease in SV (ΔSV-LRM) to predict fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients receiving laparotomy and lung protective ventilation

Exclusion Criteria:

* preoperative arrhythmia
* Severe bradycardia
* Moderate to severe valvular disease
* left ventricular ejection fraction < 50%
* Poorly controlled hypertension (systolic BP > 160 mmHg)
* Patients with renal insufficiency (creatinine > 1.5 mg/dL)
* Moderate to severe liver disease
* BMI >.30 or < 15 kg/ m2
* preexisting pulmonary disease
* FEV1 < 60% of predicted value

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: tertiary care center
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
PPV_augmented | During the last 5 second of lung recruitment maneuver
  augmented pulse pressure variation by lung recruitment maneuver
SVV_augmented | During the last 5 second of lung recruitment maneuver
  augmented stroke volume variation by lung recruitment maneuver

SECONDARY OUTCOMES:
ΔSV_LRM | During the last 5 second of lung recruitment maneuver
  The degree of reduction of stroke volume induced by lung recruitment maneuver
ΔETCO2_LRM | During the last 5 second of lung recruitment maneuver
  The degree of reduction of end tidal CO2 concentration induced by lung recruitment maneuver

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sacred Heart Hospital, Hallym University College of Medicine, Seoul, South Korea